CLINICAL TRIAL: NCT07407777
Title: Evaluation of Gut-Related Well-Being and Mood Effects of a Daily Nutritional Food Ingredient From the Co-Fermentation of Fungal Mycelium (Pleurotus Pulmonarius) and Microalgae (Chlorella Vulgaris) in Healthy Adults Experiencing Minor Gastrointestinal Discomfort: A 30-Day, Two-Arm, Open-Label Study
Brief Title: Evaluation of Gut-Related Well-Being and Mood Effects of a Daily Nutritional Food Ingredient From the Co-Fermentation of Fungal Mycelium (Pleurotus Pulmonarius) and Microalgae (Chlorella Vulgaris)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koralo GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KOR001
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Gastrointestinal Discomfort; Digestive Well Being; Gut-related Symptoms
Keywords: gut health; gastrointestinal symptoms; functional food ingredient; mood and well-being; dietary intervention

STUDY DESIGN:
Intervention Model Description: Participants are randomized into two parallel intervention arms receiving different fixed daily doses of the investigational food ingredient (high-dose and low-dose) over a 30-day period. There is no placebo or crossover; outcomes are assessed longitudinally at baseline, Day 15, and Day 30
Masking Description: Not applicable. This is an open-label study in which participants and study staff are aware of dose assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Dose (Experimental): Participants assigned to this arm will consume 600 mg per day of the investigational food ingredient (active blend) derived from the co-fermentation of Pleurotus pulmonarius mycelium and Chlorella vulgaris microalgae. The powdered product will be taken once daily for 30 days by mixing it into a beverage of the participant's choice. Gastrointestinal symptoms and mood-related outcomes will be assessed at baseline, Day 15, and Day 30 using validated self-report questionnaires.
  Interventions: Dietary Supplement: Food ingredient of oyster mushroom mycelium (Pleurotus pulmonarius) and microalgae (Chlorella vulgaris)
- High Dose (Experimental): Participants assigned to this arm will consume 4,000 mg per day of the investigational food ingredient (active blend) derived from the co-fermentation of Pleurotus pulmonarius mycelium and Chlorella vulgaris microalgae. The powdered product will be taken once daily for 30 days by mixing it into a beverage of the participant's choice. Gastrointestinal symptoms and mood-related outcomes will be assessed at baseline, Day 15, and Day 30 using validated self-report questionnaires.
  Interventions: Dietary Supplement: Food ingredient of oyster mushroom mycelium (Pleurotus pulmonarius) and microalgae (Chlorella vulgaris)

INTERVENTIONS:
Dietary Supplement: Food ingredient of oyster mushroom mycelium (Pleurotus pulmonarius) and microalgae (Chlorella vulgaris) — Food ingredient obtained from the co-fermentation of oyster mushroom mycelium (Pleurotus pulmonarius), microalgae (Chlorella vulgaris) and added bamboo fibre with flavours for better palatability

SUMMARY:
The purpose of the study is to evaluate the gut-related well-being and mood effects of a food ingredient obtained from the co-fermentation of oyster mushroom mycelium (Pleurotus pulmonarius), microalgae (Chlorella vulgaris), and bamboo fibre in healthy adults (aged 18+) experiencing minor gastrointestinal discomfort during an intervention period of 30 days. The participants will be allocated into two unbalanced groups to determine relationships between the measurable outcomes and the dose levels at three different time points: start of the study (baseline), 15 days (middle), and 30 days (end-point), during which participants will be asked to complete GSRS and POMS-2-SF questionnaire

DETAILED DESCRIPTION:
This study is a 30-day, two-arm, open-label dietary intervention designed to evaluate the effects of a daily nutritional food ingredient on gastrointestinal well-being and mood in generally healthy adults experiencing minor, non-clinical gastrointestinal discomfort. The investigational product is a powdered food ingredient derived from the co-fermentation of fungal mycelium (Pleurotus pulmonarius) and microalgae (Chlorella vulgaris), blended with bamboo fiber and flavoring components for palatability. The product is food-grade, manufactured under cGMP conditions, and supported by a self-declared GRAS safety dossier. The study will enroll a total of 80 adult participants (aged 18-65) in the United States using a fully remote, decentralized design conducted through the Alethios digital research platform.

Participants who meet eligibility criteria will be randomly assigned in an unbalanced allocation to one of two fixed-dose intervention groups: a high-dose arm receiving 4,000 mg/day of the active blend (n=50) or a low-dose arm receiving 600 mg/day (n=30). All participants will consume the assigned product once daily for 30 days by mixing the powder into a beverage of their choice. No placebo group is included, as the primary objective is to explore dose-related effects rather than to compare against no treatment. The study involves no invasive procedures, clinical visits, laboratory testing, or biological sample collection, and participants may continue their usual diet and daily activities throughout the study period.

Study outcomes will be assessed using validated, self-reported questionnaires administered electronically at three time points: baseline (Day 0), mid-intervention (Day 15), and end of study (Day 30). The primary outcome is change in gastrointestinal symptom severity, measured by the Gastrointestinal Symptom Rating Scale (GSRS). Secondary outcomes include changes in mood and psychological well-being, assessed using the Profile of Mood States-2 Short Form (POMS-2-SF), as well as changes in GSRS subscale scores. Exploratory analyses will compare effect sizes between the two dose levels to assess potential dose-response relationships. Participant burden is minimal, with an estimated total time commitment of approximately 90 minutes over the entire study.

The study is classified as minimal risk, with anticipated risks limited to mild and transient gastrointestinal symptoms or rare allergic reactions consistent with the introduction of new dietary ingredients. Safety monitoring is conducted through daily self-report check-ins and adverse event reporting within the digital platform, with automated alerts to study staff as needed. Participants may withdraw at any time without penalty. Collectively, the study is designed to generate preliminary human evidence on the safety, tolerability, and potential benefits of the investigational food ingredient for gastrointestinal comfort and overall well-being in a mildly symptomatic, otherwise healthy adult population, providing a strong scientific rationale for future research.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 years or older

Generally healthy individuals

Experience minor, non-clinical gastrointestinal discomfort at least twice per week for ≥3 months

Willing to consume the study product once daily for 30 days

Able to dissolve and consume the powdered product in a beverage

Able to read, understand, and complete electronic questionnaires in English

Access to a smartphone or computer for study participation

Provide electronic informed consent

Exclusion Criteria:

* Diagnosed gastrointestinal disease (e.g., IBS, IBD, GERD requiring medication)

Use of medications affecting gastrointestinal function or mood within the past 30 days

Initiation of new gut-, immune-, or mood-related supplements within 15 days prior to study start

Known allergy or sensitivity to study product components

Pregnancy or breastfeeding

Major chronic medical condition that could interfere with study participation or data interpretation

Participation in another interventional clinical study within the past 30 days

Inability or unwillingness to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-19 (Actual); Primary Completion 2026-05-19 (Estimated); Study Completion 2026-05-19 (Estimated)

PRIMARY OUTCOMES:
Change in Gastrointestinal Symptom Rating Scale (GSRS) Total Score | Baseline (Day 0) to Day 30
  The primary outcome is the change in gastrointestinal symptom severity as measured by the Gastrointestinal Symptom Rating Scale (GSRS). The GSRS is a validated self-report questionnaire assessing the severity of common gastrointestinal symptoms. Change in total GSRS score will be evaluated over the course of the 30-day intervention to assess the effect of the investigational food ingredient on gut-related well-being.

SECONDARY OUTCOMES:
Change in Profile of Mood States-2 Short Form (POMS-2-SF) Total Mood Disturbance Score | Baseline (Day 0) to Day 30
  The secondary outcome is the change in mood and psychological well-being as measured by the Profile of Mood States-2 Short Form (POMS-2-SF). The POMS-2-SF is a validated self-report questionnaire assessing mood states across multiple domains. Change in total mood disturbance score will be evaluated to assess the effect of the investigational food ingredient on mood and overall well-being during the intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- Alethios, Inc., San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided